CLINICAL TRIAL: NCT04449354
Title: A Study to Evaluate the HS Specific Wound Dressing HidraWear AX in the Home Setting
Brief Title: HidraWear Study for Hidradenitis Suppurativa Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HidraMed Solutions Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CE-GAX-001-01 V4
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa; Hidradenitis
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality of Life assessment (Other): HidraWear AX Garment
  Interventions: Device: HidraWear Ax

INTERVENTIONS:
Device: HidraWear Ax — An adhesive free wound dressing fixation device for people living with Hidradenitis Suppurativa (HS), Hidrawear AX, designed to make dressing changes quick and easy for subjects. The unique features of the product completely remove the use of adhesives on the skin.The body conforming garment acts as a second skin and incorporates largely perforated panels over wound affected areas, minimising skin contact and aerating the area. The main function of the perforated is to act as a retaining device for the wound pads. The garment facilitates easy insertion, removal, precise positioning and adjustment of a non- adhesive wound dressing onto the effected wound space. The perforated section of the garment sits on the outer surface of the dressing providing provisional fixation. Next, an outer patch is placed on the outside of the garment on the footprint of the dressing. Through a hook and loop mechanism the dressing is now fully secured in place.

SUMMARY:
The product, HidraWear AX (www.hidrawear.com) is and adhesive free wound dressing system for the every day home care of Hidradenitis Suppurativa (HS), a debilitating disease of the skin for which there are limited wound dressing products.

This is a study to assess the use HidraWear Ax vs current product and method of use, and to determine the impact on patients' quality of life.

DETAILED DESCRIPTION:
The objective is to evaluate the ease of use of Hidrawear AX compared to the subject's existing product use in 23 subjects with HS (Hidradenitis Suppurativa).

Secondary objectives are to evaluate if Hidrawear AX:

* Is comfortable
* Improves quality of life
* Faster to use than the subject's existing product
* Reduces dressing related pain
* Secure dressing retention

This pilot study will evaluate usability - the safety, efficacy and performance of HidraWear AX in the home setting. Quality of life, ease of use and comfort of Hidrawear AX will be assessed.

The clinical effect of the wound pad will not be assessed.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  1. Provision of signed and dated informed consent form in English.
  2. Stated willingness to comply with all study procedures and availability for the duration of the study
  3. Female, aged >18
  4. Diagnosed with Hidradenitis Suppurativa
  5. Hidradenitis Suppurativa affecting the axilla
  6. Exuding lesion that requires wound dressings

Exclusion Criteria:

* 1. Recent surgery <3 months in axilla 2. Psoriasis, Dermatitis or skin conditions/rash other than Hidradenitis Suppurativa on or near affected area 3. Pregnancy or lactation 4. Known allergic reactions to components of Hidrawear AX

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Product is designed for females
Enrollment: 16 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Duffy, Principal Investigator — Hermitage Clinic
Locations (1):
- The Hermitage Clinic, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HidraWear AX: HidraWear AX Garment
  HidraWear Ax: An adhesive free wound dressing fixation device for people living with Hidradenitis Suppurativa (HS), Hidrawear AX, designed to make dressing changes quick and easy for subjects. The unique features of the product completely remove the use of adhesives on the skin.The body conforming garment acts as a second skin and incorporates largely perforated panels over wound affected areas, minimising skin contact and aerating the area. The main function of the perforated panel is to act as a retaining device for the wound pads. The garment facilitates easy insertion, removal, precise positioning and adjustment of a non- adhesive wound dressing onto the effected wound space.
  Participants used HidraWear AX for 21 days
Period: Overall Study
Arm/Group | HidraWear AX
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | HidraWear AX
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Ireland | 16

OUTCOME MEASURES:

1. Primary Outcome: Ease of Use Day 21 vs Day 0
Description: 10 point visual analogue scale with a maximum score of 10 and a minimum score of 0. self reported . A score of 0 means the product is very easy to use, and a score of 10 means the product is very difficult to use. A lower score represents a better outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HidraWear AX
Number analyzed (Participants) | 15
score on a scale
  Day 0 | 6.47 (2.75)
  Day 21 | 0.6 (1.59)

2. Secondary Outcome: Change in Quality of Life (QoL) Measured Using the Dermatology Life Quality Index (DLQI)
Description: The Dermatology Life Quality Index (DLQI) is a ten-item questionnaire designed to measure the impact of skin diseases on patients' quality of life, focusing on symptoms, daily activities, leisure, work or school, personal relationships, and treatment. It provides a quick and quantifiable assessment, with scores ranging from 0 (no impact) to 30 (extremely large impact), facilitating the evaluation of disease severity and treatment efficacy. A lower score represents a better outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score in the DLQI Questionnaire
Arm/Group | HidraWear AX
Number analyzed (Participants) | 15
score in the DLQI Questionnaire
  Day 0 | 19.3 (5.73)
  Day 21 | 4.53 (3.93)

3. Secondary Outcome: Visual Pain Analogue Scale Day 21 vs Day 0
Description: Patient reported pain, 10 point scale, high score indicates pain. 10 point visual analogue scale with a maximum score of 10 and a minimum score of 0. self reported . A score of 0 means the patient experiences no pain, and a score of 10 means the patient experiences extreme pain. A lower score represents a better outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HidraWear AX
Number analyzed (Participants) | 15
score on a scale
  Day 0 | 5.53 (2.50)
  Day 21 | 0.80 (1.67)

4. Secondary Outcome: Time Taken to Dress Wounds
Description: 10 point visual analogue scale with a maximum score of 10 and a minimum score of 0. Self reported . A score of 0 means the product is very quick to use, and a score of 10 means the product is very time consuming to use. A lower score represents a better outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HidraWear AX
Number analyzed (Participants) | 15
score on a scale
  Day 0 | 6.93 (2.46)
  Day 21 | 0.67 (1.4)

5. Secondary Outcome: Body Image Visual Analogue Scale
Description: 10 point visual analogue scale with a maximum score of 10 and a minimum score of 0. Self reported . A score of 0 means the patient feels confident about their body image, and a score of 10 means the patient does not feel confident at all about their body image. A lower score represents a better outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HidraWear AX
Number analyzed (Participants) | 15
score on a scale
  Day 0 | 8.53 (1.92)
  Day 21 | 3.8 (2.18)

6. Secondary Outcome: Patient Comfort
Description: 10 point visual analogue scale with a maximum score of 10 and a minimum score of 0. Self reported . A score of 0 means the product is very comfortable to use and wear, and a score of 10 means the product is very uncomfortable to use and wear. A lower score represents a better outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HidraWear AX
Number analyzed (Participants) | 15
score on a scale
  Day 0 | 8.13 (1.92)
  Day 21 | 1 (1.25)

7. Secondary Outcome: Confidence in Dressing Product (Secure Retention, Leak Reduction)
Description: 10 point visual analogue scale with a maximum score of 10 and a minimum score of 0. Self reported . A score of 0 means the patient is confident in the products ability to remain in place and contain exudate, and a score of 10 indicates low confidence in products ability to remain in place or contain exudate. A lower score represents a better outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HidraWear AX
Number analyzed (Participants) | 15
score on a scale
  Day 0 | 8.4 (2.53)
  Day 21 | 1.2 (1.82)

ADVERSE EVENTS:
Time Frame: 1 year
Description: This study was for a non invasive, class one medical device. Risk assessment and mitigation in place. All-Cause Mortality was not monitored/assessed.
Arm/Group | HidraWear AX
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT04449354/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT04449354/ICF_001.pdf